CLINICAL TRIAL: NCT06384586
Title: Investigation of Dietary Supplement Liquid Shot Products on Mental Energy, Cognition (Acuity),and Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Water Street Collective (Industry)
Collaborators: HCD Research (Industry); British American Tobacco (Investments) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: CD J8855
Record Dates: First submitted 2024-04-17; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Cognition; Mental Fatigue; Mood
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo 60 ml Shot, matched in volume, taste and colour and did not contain any active ingredients. 1 shot to be consumed per session
  Interventions: Dietary Supplement: Placebo shot; Dietary Supplement: Functional energy shot
- Functional Energy shot (Experimental): 60ml functional energy shot contained a proprietary blend of caffeine, ginseng, vitamins and taurine. 1 shot to be consumed per session
  Interventions: Dietary Supplement: Placebo shot; Dietary Supplement: Functional energy shot

INTERVENTIONS:
Dietary Supplement: Placebo shot — 60ml shot served in an amber bottle and consumed after 40 minutes of baseline assessments
Dietary Supplement: Functional energy shot — 60ml shot served in an amber bottle and consumed after 40 minutes of baseline assessments

SUMMARY:
This is a single center, randomized, double blind, placebo-controlled, crossover study to determine the acute effect of a developmental dietary supplement liquid shot product on cognitive task performance and perceived effect measures related to mood and mental energy. The study will be conducted in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

MAIN INCLUSION CRITERIA:

1. Participants must be willing to abstain from alcohol, caffeine and exercise starting from the night before each session.
2. Participants that, on average, consume between 200 and 500 mgs of caffeine per day.
3. Participants that are in good physical and mental health.
4. Participants that are willing to come in-person and be within less than 6 feet of study staff for a short period of time.
5. Participants that are able to provide written informed consent to participate in the study and will have agreed to abide by the study restrictions, requirements and protocol.
6. Participants must, in the opinion of the Principal Investigator (or designee), demonstrate the ability to comprehend the informed consent form (ICF), be able to communicate well with the Investigator, understand and comply with the requirements of the study, and be judged suitable for the study.
7. Participants must be available to complete the study.
8. Participants must be willing to consume a normal-sized meal (participant responsible for obtaining or preparing the meal) at least one hour prior to the start of the study session and then fast from food and beverage consumption (except water), for one hour prior to each research session.

Exclusion Criteria:

1. Participants that are not US citizens or are residents of California.
2. Participants that have a medical condition, including but not limited to heartbeat/rhythm irregularities, past heart attacks, been diagnosed with heart disease, seizure disorder, liver condition, blood clotting disorder, endocrine-related medical diagnosis (such as diabetes, thyroid, etc.), serious health condition (i.e. cancer, etc.), blindness, gastrointestinal sensitivity/condition, depression, insomnia, anxiety, hypertension, PKU (Phenylketonuria), Celiac disease or deafness. If a participant has any other medical condition or metabolic condition that prevents them from being able to fast for one hour, they will not be allowed to participate in this study.
3. Participants that have a loss of taste or smell or are currently suffering from a virus/infection that affects their ability to taste or smell.
4. Participants that are left-handed, have dyscalculia, have paralysis which effects the upper body, or are color-blind, as this could impact their ability to complete the cognitive tasks.
5. Participants that use recreational drugs or that are currently taking medication (except for a contraceptive), or other drugs including non-prescription (over the counter) medications, pseudoephedrine, non-prescription painkillers such as paracetamol (acetaminophen), ibuprofen or aspirin.
6. Participants that are taking green tea extract or any diet medications, appetite suppressors or supplements (including, but not limited to, fitness supplements containing green tea extract and caffeine, and workout supplements that are intended to assist with weight loss (such as phentermine)).
7. Participants that are pregnant, breastfeeding (or pumping/expressing) or intend to become pregnant in the next six months.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Mental energy via Cognitive Demand Battery (CDB) Performance Index; for the functional energy shot versus placebo shot. | Change from baseline to 120 min post- shot consumption
  CDB performance index score is a comprised averaged Z scores for the principal performance measure for each of the three tasks: Rapid Visual Information Processing (RVIP) % accuracy, Serial 3s total number correct, Serial 7s total number correct. A higher score signifies performance improvement. Objective tests within Computerised Mental Performance Assessment framework tasks (COMPASS)

SECONDARY OUTCOMES:
Mental energy via Cognitive Demand Battery (CDB) Accuracy score for the functional energy shot versus placebo shot. | Change from baseline to 120 min post- shot consumption
  CDB accuracy score is a comprised averaged Z scores for the principal measures of accuracy of performance for the three tasks: Rapid Visual Information Processing (RVIP) % accuracy; Serial 3s % errors; Serial 7s % errors (the latter two were inverted so that a higher Z score related to better accuracy). A higher score signifies performance improvement.
  Objective tests within Computerised Mental Performance Assessment framework tasks (COMPASS)
Change in performance on Corsi blocks task for functional energy shot versus placebo | Change from baseline to 120 min post- shot consumption
  Objective tests within Computerised Mental Performance Assessment framework tasks (COMPASS)
Change in performance on Rapid Visual Information Processing (RVIP) for functional energy shot versus placebo | Change from baseline to 120 min post- shot consumption
  Objective tests within Computerised Mental Performance Assessment framework tasks (COMPASS)
Change in performance on Numeric working memory for functional energy shot versus placebo | Change from baseline to 120 min post- shot consumption
  Objective tests within Computerised Mental Performance Assessment framework tasks (COMPASS)
Change in performance on Serial subtraction task for functional energy shot versus placebo | Change from baseline to 120 min post- shot consumption
  Objective tests within Computerised Mental Performance Assessment framework tasks (COMPASS)
Change in Mood via Visual Analogue Scales (VAS) during Cognitive Demand Battery (CDB), for functional energy shot versus placebo | Change from baseline to 120 min post- shot consumption
  0-100 mm subjective rating scale from none to strongest feelings, within Computerised Mental Performance Assessment framework tasks (COMPASS) for mental fatigue, alert, sociable, simulated, jittery, physical energy. The minimum score is 0 and the maximum score is 100.
Change in physiological state via Profile Of Mood States (POMS) during Cognitive Demand Battery (CDB), for functional energy shot versus placebo | Change from baseline to 120 min post- shot consumption
  a 37-item inventory, the individual item scores of which are collapsed into six dimensions of mood: anger/hostility, confusion/bewilderment, depression/dejection, fatigue/inertia, tension/anxiety, and vigour/activity.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle M Niedziela, PhD, Principal Investigator — HCD Research
Locations (1):
- Schlesinger Group New Jersey, Iselin, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] O'Shea OK, Lawley N, Azzopardi A, Gutkowski A, Niedziela MM, Horn R, Kennedy DO, Adamson J. Acute beneficial effects of a functional energy shot on cognitive performance and mood states during cognitively demanding task performance: a randomized, double-blind, placebo-controlled, crossover trial. Front Nutr. 2025 Jan 9;11:1496092. doi: 10.3389/fnut.2024.1496092. eCollection 2024. PMID 39850336